CLINICAL TRIAL: NCT05168033
Title: The Effect of Motor Imagery as an Additional Tool During the Rehabilitation After Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial
Brief Title: Motor Imagery After Reconstruction of the Anterior Cruciate Ligament
Acronym: MIRACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6702021000881
Record Dates: First submitted 2021-11-09; First posted 2021-12-23 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Anterior Cruciate Ligament Rupture; Motor Imagery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery training (Experimental): In addition to classic rehabilitation the experimental group will be assigned to motor imagery training.
  This training will take place at 3 specific periods (4 weeks) during the rehabilitation process:
  MI 1: immediately postoperative; MI 2: return to run; MI 3: change of directions and cutting;
  To complete a motor imagery training session, participants of the experimental group will have to watch video clips in which rehabilitation exercises or sport specific situations will be shown. After watching, participants will have to mentally imagine they are performing these exercises themselves without actually moving. During each of the 3 motor imagery periods, subjects will be required to complete 20 sessions of 10-15 minutes each.
  Interventions: Other: Motor imagery training; Other: Classic rehabilitation
- Classic rehabilitation (Active Comparator): This group will follow the classic rehabilitation pathway after anterior cruciate ligament reconstruction.
  Interventions: Other: Classic rehabilitation

INTERVENTIONS:
Other: Motor imagery training — Mentally imagine to perform rehabilitation exercises or sport-specific tasks without generating actual motor output.
  Other Names: Mental practice
  Arms: Motor imagery training
Other: Classic rehabilitation — Classic rehabilitation after anterior cruciate ligament reconstruction focusing on regaining mobility, stability and strength of the knee joint and return to sport.

SUMMARY:
The primary aim of this study is to investigate the effect of motor imagery training as an additional tool in the rehabilitation after anterior cruciate ligament reconstruction (ACLR). Therefore, ACLR patients will be recruited and randomly assigned into one of following groups:

* Experimental group: Classic rehabilitation + Motor imagery training
* Control group: Classic rehabilitation

Both, the control and experimental group, will be submitted to a routine physiotherapy program after ACLR. In addition, the intervention group will be exposed to motor imagery training at three different time periods during the rehabilitation process (MI 1: immediately postoperative; MI 2: return to run; MI 3: change of direction). All participants will be invited for a preoperative screening, several postoperative screenings at 4-week time intervals and a final return to sport screening. At these test moments, participants will be subjected to a specific test battery consisting of subjective and objective clinical parameters. The subjective outcomes imply the patient's perception of pain and discomfort, level of participation, psychosocial well-being and overall quality of life. The objective clinical outcome measures relate to knee mobility and muscle strength, level of functioning/performance capacity and the detection of brain areas and networks involved in the processes of anxiety and worrying using EEG.

DETAILED DESCRIPTION:
To investigate the effect of motor imagery training in addition to classical rehabilitation after anterior cruciate ligament reconstruction, a randomized study with prospective follow-up will be set up in an adult population of both male and female subjects.

After recruitment, patients who are eligible to participate in the study will be randomly assigned to either the experimental group or the control group. Both groups will follow the standard rehabilitation program after anterior cruciate ligament reconstruction to promote mobility, strength, proprioception, stability and return to sport.

For the participants in the experimental group, motor imagery training will be included in the rehabilitation program, organized into 3 specific periods (4 weeks) during the rehabilitation process.

* MI 1: immediately postoperative (0-4w postop)
* MI 2: return to run (8-12w postop)
* MI 3: return to cutting and directional changes (16-20w postop)

These MI training sessions (MITS) will consist of watching video clips in which the subjects will be shown rehabilitation exercises or sport-specific situations. After watching, participants will have to mentally imagine they are performing these exercises themselves, without actually moving. It is important that subjects concentrate on all muscular, sensorimotor and proprioceptive sensations as they would occur during the effective performance of the exercise or task. During each of the 3 motor imagery periods, subjects will be required to complete 20 sessions of 10-15 minutes each.

Participants from the experimental group will be subjected to a specific test battery preoperatively and before and after each motor imagery training period, tailored to the stage of the rehabilitation process. Control group participants will also be subjected to this specific test battery at similar times in the rehabilitation process (preoperative, 0w, 4w, 8w, 12w, 16w, 20w and RTS testing).

Finally, all participants (experimental group + control group) will be contacted by telephone at 3 months and 1 year after the last screening to ask them about the type of sport they practice, at which level they practice this sport, how much confidence they have in their operated knee during sports and any new injuries.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament reconstruction
* Rehabilitation at the sports physiotherapy department of the Ghent University Hospital

Exclusion Criteria:

* Neurological disorders or diseases that could affect motor imagery training
* Musculoskeletal or cognitive disorders that interfere with the normal function of the lower extremities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - Questionnaire | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  Assess the patients opinion about their knee and associated problems. Each item is given a score between 0 and 4, then the total score is converted to a scale of 0-100. A higher score indicates less disfunction.
ACL-Return to sport after injury (ACL-RSI) - Questionnaire | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  This questionnaire consists of 12 questions divided into three main sections: athletes' emotion, confidence, and risk assessment when returning to sport after an ACL injury and/or reconstructive surgery.
  Each item is given a score between 0 and 100, after which the total score is converted to a scale of 0-100. A lower score indicates more concerns about return to sport.
Visual Analogue Scale (VAS) - Questionnaire | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  A validated, subjective measure for acute and chronic pain (0-100). A higher score indicates more pain.
Knee confidence - Questionnaire | From preoperative screening (1 week before surgery) until end of follow up (15 months postoperative)
  To evaluate the confidence of patients in their operated knee, expressed as a percentage relative to the nonoperated side (0-100%). A lower score indicates less confidence.
Limb circumference | From preoperative screening (1 week before surgery) until 4 weeks postoperative
  Knee effusion is measured by a tape measure at 2 different points on the thigh (5 cm and 15 cm above the patella).
Knee Flexion and Extension Range of Motion | From preoperative screening (1 week before surgery) until 4 weeks postoperative
  Using a goniometer, knee flexion and extension range of motion of the knee joint will be measured.
Quadriceps muscle strength | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  Using a handheld dynamometer the strenght of the quadriceps muscle will be measured.
Balance | From 8 weeks postoperative until return to sport screening (28 weeks postoperative)
  Dynamic balance will be measured using the Y-balance test - lower quadrant
Hop tests | From 16 weeks postoperative until return to sport screening (28 weeks postoperative)
  Single leg hop for distance, vertical jump and side hop. These tests will compare the affected and non-affected side (Limb Symmetry Index) in the context of return to sport readiness.
Change in movement quality | Respectively from 8, 12 and 24 weeks postoperative until return to sport screening (28 weeks postoperative)
  Lateral step down, drop vertical jump and a cutting maneuver task are assessed for movement quality using a 2D video camera setup.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) - Questionnaire | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  This questionnaire consists of 16 questions and evaluates the extent to which patients are concerned
  Each item is given a score between 1 and 5. The total scores range from 16 to 80 with higher scores indicative of higher levels of trait worry.
Tampa scale of Kinesiophobia (TSK) - Questionnaire | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  This questionnaire consists of 17 questions and evaluates the extent to which patients experience kinsiophobia.
  Each item is given a score between 0 and 4. A higher score indicates more kinesiophobia.
Resting state brain activity | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  Electroencephalography (EEG) will be recorded from 128 Sn surface electrodes using an electrode cap during 5 minutes of sitting on a chair. Spectral power will be analyzed.
Event-related potentials | From preoperative screening (1 week before surgery) until return to sport screening (28 weeks postoperative)
  Electroencephalography (EEG) will be recorded from 128 Sn surface electrodes using an electrode cap during 2x5 minutes of watching videoclips. Spectral power will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, Ghent University
Locations (1):
- Ghent University, Department of Rehabilitation Sciences, Ghent, Belgium